CLINICAL TRIAL: NCT02526017
Title: A Phase 1a/1b Study of Cabiralizumab in Combination With Nivolumab in Patients With Selected Advanced Cancers
Brief Title: Study of Cabiralizumab in Combination With Nivolumab in Patients With Selected Advanced Cancers
Acronym: FPA008-003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FPA008-003
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumors; Head and Neck Cancer; Pancreatic Cancer; Ovarian Cancer; Renal Cell Carcinoma; Malignant Glioma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell; Glioma; Carcinoma, Non-Small-Cell Lung | interventions — cabiralizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1a Monotherapy Dose Escalation (Experimental): Cabiralizumab administered at 2 mg/kg every 2 weeks (Q2W), 4 mg/kg Q2W and 6 mg/kg Q2W in participants with any solid tumor.
  Interventions: Biological: Cabiralizumab
- Phase 1a Combination Therapy Dose Escalation (Experimental): Nivolumab 3 mg/kg Q2W + cabiralizumab at the following doses: 1 mg/kg, 2 mg/kg, 4 mg/kg, and 6 mg/kg Q2W. Also nivolumab 3 mg/kg + cabiralizumab 4 mg/kg every 3 weeks (Q3W). Participants with any solid tumor.
  Interventions: Biological: Cabiralizumab; Biological: Nivolumab
- Phase 1b Combination Therapy Dose Expansion (Experimental): The expansion phase would use the recommended dose determined in Phase 1a: cabiralizumab 4 mg/kg + nivolumab 3 mg/kg Q2W. Participants are enrolled for the following advanced cancer types: non-small cell lung cancer (anti-programmed cell death 1 [PD1] targeted drug naïve), non-small cell lung cancer (prior treatment with anti-PD-1), pancreatic cancer, ovarian cancer, renal cell cancer, glioblastoma, and melanoma.
  Interventions: Biological: Cabiralizumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Cabiralizumab — Solution for IV administration
  Other Names: Anti-colony stimulating factor-1 receptor (Anti-CSF-1R); FPA008
Biological: Nivolumab — Solution for IV administration
  Other Names: OPDIVO®; MDX-1106; BMS-936558
  Arms: Phase 1a Combination Therapy Dose Escalation; Phase 1b Combination Therapy Dose Expansion

SUMMARY:
Phase 1a/1b does-escalation study of cabiralizumab alone and with nivolumab in advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase 1a/b single-arm, open-label study to evaluate safety, tolerability, pharmacokinetics (PK), and clinical benefit of cabiralizumab in combination with nivolumab in patients with selected advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have at least one measurable lesion at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
* Patients must have had progressive disease on, after, or refused, appropriate approved therapy for their tumor type.
* Patients must have histologically or cytologically confirmed solid tumor that is locally recurrent or metastatic and has progressed following standard treatment or is not appropriate for standard treatment
* Understand and sign an Institutional review board/Independent ethics committee (IRB/IEC)-approved informed consent form (ICF) prior to any study-specific evaluation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Current or history of clinically significant muscle disorders (e.g., myositis), recent unresolved muscle injury, or any condition known to elevate serum creatine kinase (CK) levels
* Decreased cardiac function with New York Heart Association (NYHA) > Class 2
* Uncontrolled or significant heart disorder such as unstable angina
* Significant abnormalities on electrocardiogram (ECG) at screening. Fridericia's correction formula for QT interval (QTcF) > 450 msec for males or > 470 msec for females at screening
* History of anti-drug antibodies, severe allergic, anaphylactic, or other infusion-related reaction to a previous biologic agent
* Positive test for latent tuberculosis (TB) at screening (Quantiferon test) or evidence of active TB
* Patients with abnormal serum chemistry values, which in the opinion of the Investigator is considered to be clinically significant, will be excluded from the study
* Lack of peripheral venous or central venous access or any condition that would interfere with drug administration or collection of study samples
* Any uncontrolled medical condition or psychiatric disorder which, in the opinion of the Investigator, would pose a risk to patient safety or interfere with study participation or interpretation of individual patient results
* Pregnant or breastfeeding
* Current unresolved infection or history of chronic, active, clinically significant infection (viral, bacterial, fungal, or other) which, in the opinion of the Investigator, would preclude the patient from exposure to a biologic agent or pose a risk to patient safety
* Prior exposure to any colony stimulating factor 1 receptor (CSF1R) pathway inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Lead, Study Director — Five Prime Therapeutics, Inc.
Locations (39):
- United States (39):
  - Scottsdale Healthcare Hospitals DBA Honor Health, Scottsdale, Arizona
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Norris Comprehensive Cancer Center, University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Center, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - UCLA Hematology/Oncology- Santa Monica, Santa Monica, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Health Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allina Health, Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, William M. Cooper Ambulatory Pavilion of the Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Medical University of South Carolina, Charleston, South Carolina
  - Henry-Joyce Cancer Clinic, Vanderbilt-Ingram Cancer Center,, Nashville, Tennessee
  - Baylor Charles A. Sammons Cancer Center, Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Mischer Neuroscience Associates, The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy & Research Center, University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included a Phase 1a dose escalation and a Phase 1b dose expansion. The dose escalation phase consisted of cabiralizumab monotherapy cohorts and cohorts of cabiralizumab in combination with nivolumab. All dose escalation decisions were based on assessment of dose-limiting toxicity (DLT), overall safety, and tolerability. Enrollment in Phase 1b expansion began after a recommended dose had been identified in Phase 1a.
Pre-assignment Details: The primary objective of the study was to assess the safety and tolerability of cabiralizumab alone and in combination with nivolumab. Accordingly, the safety results are grouped by patients who received the same dose and schedule of both medications. The co-primary objective for the Phase 1b portion was to evaluate the clinical benefit. Accordingly, the efficacy results from Phase 1b are reported by tumor types.
Groups:
- Phase 1a: Cabiralizumab 2 mg/kg Q2W: Participants received 2 mg/kg cabiralizumab administered intravenously (IV) once every 2 weeks (Q2W) until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 4 mg/kg Q2W: Participants received 4 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 6 mg/kg Q2W: Participants received 6 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 1 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 2 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W; Phase 1b: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 6 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W: Participants received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV every 3 weeks (Q3W) until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
Period: Overall Study
Arm/Group | Phase 1a: Cabiralizumab 2 mg/kg Q2W | Phase 1a: Cabiralizumab 4 mg/kg Q2W | Phase 1a: Cabiralizumab 6 mg/kg Q2W | Phase 1a: Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W | Phase 1b: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W
Started | 3 | 10 | 11 | 4 | 4 | 3 | 6 | 10 | 262
Received Study Treatment | 3 | 10 | 11 | 4 | 3 | 3 | 6 | 10 | 262
Completed | 3 | 10 | 11 | 4 | 3 | 3 | 6 | 10 | 262
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrew Consent Before Receiving Study Treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1a: Cabiralizumab 2 mg/kg: Participants received 2 mg/kg cabiralizumab administered intravenously (IV) once every 2 weeks (Q2W) until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 4 mg/kg: Participants received 4 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 6 mg/kg: Participants received 6 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Total: Total of all reporting groups
Arm/Group | Phase 1a: Cabiralizumab 2 mg/kg | Phase 1a: Cabiralizumab 4 mg/kg | Phase 1a: Cabiralizumab 6 mg/kg | Phase 1a: Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W | Phase 1b: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Total
Number analyzed (Participants) | 3 | 10 | 11 | 4 | 3 | 3 | 6 | 10 | 262 | 312
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 5 | 1 | 0 | 1 | 2 | 4 | 141 | 159
  >=65 years | 3 | 5 | 6 | 3 | 3 | 2 | 4 | 6 | 121 | 153
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 3 | 2 | 1 | 2 | 4 | 6 | 125 | 151
  Male | 1 | 4 | 8 | 2 | 2 | 1 | 2 | 4 | 137 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 22 | 27
  Not Hispanic or Latino | 1 | 10 | 11 | 2 | 3 | 2 | 6 | 10 | 231 | 276
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 17 | 18
  Native Hawaiian / Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 12 | 13
  White | 3 | 10 | 10 | 4 | 3 | 3 | 5 | 10 | 219 | 267
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 13
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Grade 3 or Grade 4 Adverse Events (AEs) and Laboratory Abnormalities Defined as Dose Limiting Toxicities (DLT) (Phase 1a)
Description: A DLT was defined as a study drug-related ≥ Grade 3 AE (using National Cancer Institute Common Terminology Criteria for Adverse Events v 4.03) occurring during the first 28-days, excluding Grade 3 tumor flare (defined as local pain, irritation, or rash localized at sites of known or suspected tumor), rash, immune-related adverse event (irAE) that resolved to ≤ Grade 1 by 14 days or a transient (resolving within 6 hours of onset) Grade 3 infusion-related AE. Any recurrence of Grade 3 rash, irAE or infusion-related AE was considered a DLT.
  The protocol was amended such that in the absence of clinical symptoms and other accompanying changes in bilirubin or alanine aminotransferase (ALT), serum elevation of aspartate aminotransferase (AST)/ALT > 12 × upper limit of normal (ULN) and ≤ 20 × ULN that lasted for < 7 days and serum elevation of creatine kinase (CK) and/or lactate dehydrogenase (LDH) > 15 × ULN and ≤ 20 × ULN that lasted for < 7 days were not considered DLTs.
Time Frame: 28 days
Population: Participants enrolled in the dose escalation phase who received at least 2 doses of study drug during the 28-day evaluation interval or who discontinued study treatment for drug-related adverse events before receiving 2 doses of study drug were considered evaluable for DLT determination.
Measure: Count of Participants; unit: Participants
Groups:
- Cabiralizumab 2 mg/kg Q2W: Participants received 2 mg/kg cabiralizumab administered intravenously (IV) once every 2 weeks (Q2W).
- Cabiralizumab 4 mg/kg Q2W: Participants received 4 mg/kg cabiralizumab IV Q2W
- Cabiralizumab 6 mg/kg Q2W: Participants received 6 mg/kg cabiralizumab IV Q2W.
- Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 1 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W.
- Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 2 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W.
- Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 6 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W.
Arm/Group | Cabiralizumab 2 mg/kg Q2W | Cabiralizumab 4 mg/kg Q2W | Cabiralizumab 6 mg/kg Q2W | Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W
Number analyzed (Participants) | 3 | 10 | 11 | 4 | 3 | 3 | 6
Participants
  Grade 3 CK increase | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 AST increase | 0 | 2 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Recommended Dose (RD) of Cabiralizumab in Combination With Nivolumab (Phase 1a)
Description: Using both the incidence of dose limiting toxicities (first 28 days on therapy) as well as overall tolerability and toxicities observed beyond 28 days, the RD was chosen as 4 mg/kg of cabiralizumab + 3 mg/kg nivolumab every 2 weeks to be the dose used in the Phase 1b (dose expansion). No maximum tolerated dose was identified.
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: mg/kg Q2W
Groups:
- Overall Phase 1a Dose Escalation: Participants received escalating doses of cabiralizumab monotherapy or cabiralizumab in combination with nivolumab.
Arm/Group | Overall Phase 1a Dose Escalation
Number analyzed (Participants) | 40
mg/kg Q2W | 4

3. Primary Outcome: Safety: Number of Participants With Adverse Events and Serious Adverse Events (Phase 1a and 1b)
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation, patient-administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or causes prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Was an important medical event that may jeopardize the patient or may require intervention (e.g., medical, surgical) to prevent one of the other serious outcomes listed in the definition above.
Time Frame: From first dose of study drug up to 100 days after last dose. Median (range) duration of exposure was 6 (2-32) weeks in the monotherapy cohorts and 8 (2-108) weeks for cabiralizumab and 8 (2-156) weeks for nivolumab in the combination groups.
Population: All participants who received at least 1 dose of cabiralizumab and/or nivolumab. Safety results are grouped by participants who received the same treatment regimen.
Measure: Count of Participants; unit: Participants
Groups:
- Cabiralizumab 2 mg/kg Q2W: Participants received 2 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg Q2W: Participants received 4 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 6 mg/kg Q2W: Participants received 6 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 1 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 2 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 6 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W: Participants received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV every 3 weeks (Q3W) until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
Arm/Group | Cabiralizumab 2 mg/kg Q2W | Cabiralizumab 4 mg/kg Q2W | Cabiralizumab 6 mg/kg Q2W | Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W
Number analyzed (Participants) | 3 | 10 | 11 | 4 | 3 | 265 | 6 | 10
Participants
  Any adverse event | 2 | 10 | 10 | 4 | 3 | 264 | 6 | 10
  Serious adverse events | 1 | 1 | 6 | 2 | 1 | 138 | 3 | 5

4. Primary Outcome: Safety: Number of Participants With Treatment Discontinuations, Modifications, or Interruptions Due to Adverse Events (Phase 1b)
Description: Safety: In the Phase 1b only, the incidence of treatment discontinuations, modifications, and interruptions due to adverse events.
Time Frame: From first dose of study drug up to last dose; median (range) duration of exposure was 8 (2-108) weeks for cabiralizumab and 8 (2-156) weeks for nivolumab.
Population: All participants who received at least 1 dose of cabiralizumab and/or nivolumab at the RD of 4 mg/kg cabiralizumab + 3 mg/kg nivolumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W
Number analyzed (Participants) | 265
Participants
  Cabiralizumab infusion interruptions | 0
  Cabiralizumab infusion modifications | 12
  Nivolumab infusion interruptions | 4
  Nivolumab infusion modifications | 8
  AEs leading to discontinuation of cabiralizumab or nivolumab | 54

5. Primary Outcome: Efficacy: Objective Response Rate - Investigator Assessment (Phase 1b)
Description: Objective response rate (ORR) is defined as the percentage of participants with confirmed responses of either complete response (CR) or partial response (PR). Response was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 by investigator review.
  Complete Response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumor response was assessed every 8 weeks from first dose for the first 12 months and then every 12 weeks thereafter until end of treatment; maximum duration of treatment was 156 weeks.
Population: Response-evaluable population based on investigator assessment included all participants who had a measurable lesion at baseline and had at least 1 post-baseline tumor assessment, or clinical progression, or death.
  Efficacy endpoints were specified to be analyzed by disease type for Phase 1b participants only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve): Participants with non-small cell lung cancer (NSCLC) with no prior exposure to any programmed cell death 1 (PD-1) pathway targeting drug (PD-1 naïve) received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant): Participants with NSCLC with de novo or acquired resistance to an anti-PD-1 targeting drug (PD-1 resistant) received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN: Participants with squamous cell carcinoma of the head and neck (SCCHN) received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer: Participants with pancreatic cancer received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer: Participants with advanced ovarian cancer received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC: Participants with renal cell carcinoma (RCC) received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Malignant Glioma: Participants with malignant glioma (GBM) received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma: Participants with melanoma received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
Arm/Group | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Malignant Glioma | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma
Number analyzed (Participants) | 29 | 31 | 29 | 68 | 30 | 30 | 30 | 11
percentage of participants | 6.9 [0.8 to 22.8] | 3.2 [0.1 to 16.7] | 13.8 [3.9 to 31.7] | 5.9 [1.6 to 14.4] | 13.3 [3.8 to 30.7] | 6.7 [0.8 to 22.1] | 0 [0.0 to 11.6] | 9.1 [0.2 to 41.3]

6. Secondary Outcome: Efficacy: Overall Survival (Phase 1b)
Description: Overall survival (OS) was defined as the time from first dose of study drug to death due to any cause. OS was calculated using the Kaplan-Meier method.
  Participants who did not die while on study were censored on the date they were last known to be alive.
Time Frame: From first dose of study drug up to the end of study; maximum time on study in Phase 1b was 35.9 months.
Population: All treated participants in Phase 1b; Efficacy endpoints were specified to be analyzed by disease type for phase 1b participants only.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve): Participants with NSCLC with no prior exposure to any PD-1 pathway targeting drug (PD-1 naïve) received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN: Participants with SCCHN received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC: Participants with RCC received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: GBM: Participants with malignant glioma received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
Arm/Group | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: GBM | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma
Number analyzed (Participants) | 30 | 31 | 30 | 68 | 31 | 30 | 30 | 11
months | 12.3 [6.1 to 19.1] | 4.7 [2.6 to 10.3] | 6.4 [3.4 to NA] — Could not be estimated due to the low number of events | 5.6 [4.0 to 8.0] | 13.9 [6.9 to 16.4] | NA [16.8 to NA] — Could not be estimated due to the low number of events | 8.1 [5.7 to 12.8] | 5.3 [1.1 to 24.8]

7. Secondary Outcome: Efficacy: Overall Survival (OS) at One Year (Phase 1b)
Description: Overall survival at one-year is defined as the percentage of participants who were alive one year after receiving their first dose of study drug.
Time Frame: 52 weeks
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: GBM | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma
Number analyzed (Participants) | 30 | 31 | 30 | 68 | 31 | 30 | 30 | 11
percentage of participants | 51.1 [31.7 to 67.6] | 29.2 [13.7 to 46.6] | 42.5 [23.0 to 60.7] | 27.2 [15.8 to 39.9] | 52.9 [30.6 to 71.0] | 77.8 [57.1 to 89.3] | 35.0 [16.2 to 54.6] | 36.4 [9.0 to 65.4]

8. Secondary Outcome: Efficacy: Duration of Response (Phase 1b)
Description: Duration of response (DOR) is defined as the time from the date of the first documentation of confirmed response (CR or PR) to the first objective documentation of progressive disease (PD) per RECIST v1.1 per Investigator assessment or to death due to any cause in the absence of documented PD.
  DOR was analyzed using Kaplan-Meier methods. Participants who discontinued from the study, did not die or have disease progression, or who received new anticancer therapy were censored on the date of last evaluable assessment prior to initiation of subsequent therapy. Participants with no evaluable baseline or post-baseline assessments were censored on the date of first dose.
  Progressive Disease (PD): The appearance of one or more new lesions or at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first dose of study drug up to the end of study; maximum time on study in Phase 1b was 35.9 months.
Population: Phase 1b response-evaluable population based on investigator assessment with documented CR or PR.
  Efficacy endpoints were specified to be analyzed by disease type for Phase 1b participants only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Malignant Glioma | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma
Number analyzed (Participants) | 2 | 1 | 4 | 4 | 4 | 2 | 0 | 1
months | 8.9 [7.6 to 10.2] | 16.2 [NA to NA] — Could not be calculated for a sample size of 1 | NA [NA to NA] — Could not be calculated due to the low number of events | 12.7 [8.0 to 16.4] | 7.3 [3.8 to NA] — Could not be calculated due to the low number of events | NA [3.7 to NA] — Could not be calculated due to the low number of events |  | NA [NA to NA] — Median could not be calculated due to the low number of events; 95% confidence interval could not be calculated or a sample size of 1

9. Secondary Outcome: Efficacy: Progression Free Survival (Phase 1b)
Description: Progression-free survival (PFS) was defined as as the time from the first dose to the first objectively documented disease progression per RECIST v1.1 per Investigator assessment or death due to any cause in the absence of documented progressive disease (PD). PFS was analyzed using Kaplan-Meier methods. Participants who discontinued from the study, did not die or have disease progression, or who received new anticancer therapy were censored on the date of last evaluable assessment prior to initiation of subsequent therapy. Participants with no evaluable baseline or post-baseline assessments were censored on the date of first dose.
Time Frame: From first dose of study drug up to the end of study; maximum time on study in phase 1b was 35.9 months.
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: GBM | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma
Number analyzed (Participants) | 30 | 31 | 30 | 68 | 31 | 30 | 30 | 11
months | 2.8 [1.7 to 4.8] | 1.9 [1.7 to 3.4] | 1.8 [1.4 to 3.8] | 1.7 [1.6 to 1.9] | 2.0 [1.7 to 3.6] | 2.9 [1.8 to 5.5] | 1.8 [1.3 to 3.4] | 1.8 [1.1 to 4.9]

10. Secondary Outcome: Efficacy: Objective Response Rate - Central Review Assessment (Phase 1b)
Description: Objective response rate is defined as the percentage of participants with confirmed responses of either complete response (CR) or partial response (PR). Response was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 by independent central review.
  Complete Response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 5
Population: Response-evaluable population based on central review assessment included all participants who had at least 1 post-baseline tumor assessment, or clinical progression, or death.
  Efficacy endpoints were specified to be analyzed by disease type for phase 1b participants only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: GBM | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma
Number analyzed (Participants) | 29 | 31 | 28 | 67 | 30 | 30 | 30 | 11
percentage of participants | 3.4 [0.1 to 17.8] | 0 [0.0 to 11.2] | 10.7 [2.3 to 28.2] | 6.0 [1.7 to 14.6] | 6.7 [0.8 to 22.1] | 16.7 [5.6 to 34.7] | 0 [0.0 to 11.6] | 9.1 [0.2 to 41.3]

11. Secondary Outcome: Pharmacokinetics (PK) of Cabiralizumab: Area Under the Concentration Curve From Time Zero to Time of Last Quantifiable Concentration (AUC0-t) Normalized by Dose (Phase 1a and 1b)
Description: Cabiralizumab serum concentration was determined using a validated enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Cycles 1 and 8, Day 1 predose, and at 0.25, 4, 24, 72, 168, and 336 hours after the end of infusion.
Population: The PK evaluable population included participants who received at least 1 dose of cabiralizumab, had at least 1 available serum concentration data, and adequate PK assessments which could be used to reliably derive at least 1 PK parameter. Not all participants completed 8 cycles.
  PK data are reported by treatment regimen for Phase 1a participants and by disease type for Phase 1b participants.
Measure: Mean (Standard Deviation); unit: days*µg/mL/mg
Groups:
- Cabiralizumab 2 mg/kg Q2W: Participants with any solid tumor received 2 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg Q2W: Participants with any solid tumor received 4 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 6 mg/kg Q2W: Participants with any solid tumor received 6 mg/kg cabiralizumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W: Participants with any solid tumor received 1 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W: Participants with any solid tumor received 2 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Participants with any solid tumor received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W: Participants with any solid tumor received 6 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W: Participants with any solid tumor received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q3W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
Arm/Group | Cabiralizumab 2 mg/kg Q2W | Cabiralizumab 4 mg/kg Q2W | Cabiralizumab 6 mg/kg Q2W | Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: GBM | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma
Number analyzed (Participants) | 3 | 10 | 9 | 4 | 3 | 3 | 5 | 10 | 27 | 29 | 27 | 63 | 30 | 30 | 26 | 10
days*µg/mL/mg
  Cycle 1 | 1.26 (0.588) | 1.70 (0.444) | 1.84 (0.684) | 0.66 (0.346) | 1.22 (0.970) | 1.66 (0.737) | 2.14 (0.509) | 1.75 (0.982) | 1.74 (0.769) | 1.46 (0.562) | 1.42 (0.404) | 1.52 (0.494) | 1.95 (0.753) | 1.31 (0.460) | 2.09 (0.733) | 1.48 (0.587)
  Cycle 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 4 | 8 | 8 | 4 | 8 | 6 | 4
  Cycle 8 |  |  |  |  |  |  | 3.65 (0.696) |  | 2.83 (1.602) | 3.52 (1.290) | 2.63 (1.128) | 2.32 (0.694) | 2.69 (1.307) | 2.67 (2.120) | 4.69 (2.058) | 4.43 (1.126)

12. Secondary Outcome: PK of Cabiralizumab: Maximum Observed Concentration (Cmax) and Minimum Observed Concentration (Cmin)
Description: Cabiralizumab serum concentration was determined using a validated enzyme-linked immunosorbent assay method.
  Cmax is the maximum observed serum concentration of cabiralizumab during the dosing period.
  Cmin is the minimum observed serum concentration of cabiralizumab during a dosing interval (excluding pre-dose concentration before the first dose).
Time Frame: Cycles 1 and 8, Day 1 predose, and at 0.25, 4, 24, 72, 168, and 336 hours after the end of infusion.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Cabiralizumab 2 mg/kg Q2W | Cabiralizumab 4 mg/kg Q2W | Cabiralizumab 6 mg/kg Q2W | Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Naïve) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: NSCLC (PD-1 Resistant) | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: SCCHN | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Pancreatic Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Ovarian Cancer | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: RCC | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: GBM | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Melanoma
Number analyzed (Participants) | 3 | 10 | 9 | 4 | 3 | 3 | 5 | 10 | 27 | 29 | 27 | 63 | 30 | 30 | 26 | 10
µg/mL
  Cmax Cycle 1 | 52.11 (10.663) | 104.82 (21.543) | 142.83 (38.528) | 21.93 (7.651) | 49.00 (17.314) | 104.47 (6.890) | 124.36 (8.825) | 85.45 (16.750) | 93.41 (25.708) | 93.69 (23.406) | 83.01 (37.646) | 81.40 (17.451) | 102.62 (23.863) | 87.42 (22.209) | 103.09 (18.816) | 92.06 (13.515)
  Cmin Cycle 1 | 2.68 (2.223) | 28.61 (17.127) | 37.08 (18.490) | 3.29 (4.414) | 3.96 (2.711) | 25.57 (16.098) | 28.76 (5.307) | 10.34 (8.351) | 16.22 (10.176) | 17.82 (10.054) | 13.65 (6.959) | 15.45 (9.663) | 25.07 (12.496) | 14.19 (9.111) | 31.96 (16.282) | 17.75 (12.316)
  Cmax Cycle 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 4 | 8 | 8 | 4 | 8 | 6 | 4
  Cmax Cycle 8 |  |  |  |  |  |  | 187.27 (63.438) |  | 126.01 (39.937) | 142.85 (44.856) | 97.24 (25.252) | 108.76 (24.249) | 130.17 (29.845) | 121.06 (40.392) | 167.66 (47.960) | 164.47 (15.283)
  Cmin Cycle 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 7 | 4 | 8 | 8 | 4 | 8 | 6 | 4
  Cmin Cycle 8 |  |  |  |  |  |  | 109.66 (58.420) |  | 38.79 (20.999) | 52.26 (6.642) | 37.05 (13.674) | 40.63 (11.189) | 36.95 (15.291) | 40.15 (16.612) | 85.33 (30.039) | 82.00 (12.572)

13. Secondary Outcome: Immunogenicity of Cabiralizumab: Number of Participants With Anti-Cabiralizumab Antibodies (Phase 1a and 1b)
Description: Anti-drug antibodies (ADA) to cabiralizumab in serum were measured by a validated bridging electrochemiluminescence assay (ECLA).
  Baseline ADA Positive is defined as participants who had a baseline ADA sample which tested as positive for an anti-drug antibody against cabiralizumab; Post baseline ADA Positive is defined as participants that either had 1) an ADA detected (positive seroconversion) sample in a participant for whom ADA was not detected at baseline, or (2) an ADA detected sample with ADA titer at least 4-fold or greater than the baseline positive titer; Post baseline ADA Negative: Participants who never reported an ADA-positive sample after the initiation of treatment.
Time Frame: Blood samples were collected before the infusion on Cycles 1 (Baseline), 2, 3, 4, 5, 9, 13, and 21, and at 28 days and 100 days after the end of treatment
Population: All participants who received at least 1 dose of cabiralizumab and had available ADA data at baseline and post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabiralizumab 2 mg/kg Q2W | Cabiralizumab 4 mg/kg Q2W | Cabiralizumab 6 mg/kg Q2W | Cabiralizumab 1 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W
Number analyzed (Participants) | 3 | 10 | 11 | 4 | 3 | 263 | 6 | 10
Participants
  Baseline cabiralizumab ADA-positive | 0 | 1 | 0 | 0 | 0 | 9 | 0 | 1
  Baseline cabiralizumab ADA-negative | 3 | 9 | 11 | 4 | 3 | 254 | 6 | 9
  Cabiralizumab ADA-positive: number analyzed (Participants) | 3 | 8 | 10 | 3 | 3 | 249 | 6 | 9
  Cabiralizumab ADA-positive | 0 | 1 | 0 | 0 | 0 | 26 | 0 | 3
  Cabiralizumab ADA-negative: number analyzed (Participants) | 3 | 8 | 10 | 3 | 3 | 249 | 6 | 9
  Cabiralizumab ADA-negative | 3 | 7 | 10 | 3 | 3 | 223 | 6 | 6

14. Secondary Outcome: Immunogenicity of Nivolumab: Number of Participants With Anti-Nivolumab Antibodies (Phase 1a and 1b)
Description: Anti-drug antibodies (ADA) to nivolumab in serum were measured by a validated electrochemiluminescence assay.
  Baseline ADA Positive is defined as participants who had a baseline ADA sample which tested as positive for an anti-drug antibody against cabiralizumab; Post baseline ADA Positive is defined as participants that either had 1) an ADA detected (positive seroconversion) sample in a participant for whom ADA was not detected at baseline, or (2) an ADA detected sample with ADA titer at least 4-fold or greater than the baseline positive titer; Post baseline ADA Negative: Participants who never reported an ADA-positive sample after the initiation of treatment.
Time Frame: as for outcome 13
Population: All participants who received at least 1 dose of nivolumab and had available ADA data at baseline and post-baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Cabiralizumab 1mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 1 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
Arm/Group | Cabiralizumab 1mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W | Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W
Number analyzed (Participants) | 4 | 3 | 261 | 6 | 10
Participants
  Baseline nivolumab ADA-positive | 0 | 0 | 26 | 0 | 2
  Baseline nivolumab ADA-negative | 4 | 3 | 235 | 6 | 8
  Nivolumab ADA-positive: number analyzed (Participants) | 3 | 3 | 249 | 6 | 9
  Nivolumab ADA-positive | 1 | 0 | 57 | 1 | 3
  Nivolumab ADA-negative: number analyzed (Participants) | 3 | 3 | 249 | 6 | 9
  Nivolumab ADA-negative | 2 | 3 | 192 | 5 | 6

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 100 days after last dose. Median (range) duration of exposure was 6 (2-32) weeks in the monotherapy cohorts and 8 (2-108) weeks for cabiralizumab and 8 (2-156) weeks for nivolumab in the combination groups.
Description: All participants who received at least 1 dose of cabiralizumab and/or nivolumab. Safety results are grouped by participants who received the same treatment regimen.
Groups:
- Phase 1a: Cabiralizumab 2 mg/kg Q2W: Participants received 2 mg/kg cabiralizumab IV once every 2 weeks (Q2W) until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a: Cabiralizumab 1mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 1 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
- Phase 1a+1b: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W: Participants received 4 mg/kg cabiralizumab IV and 3 mg/kg nivolumab IV Q2W until disease progression, unacceptable toxicity, or other reason for treatment discontinuation.
Arm/Group | Phase 1a: Cabiralizumab 2 mg/kg Q2W | Phase 1a: Cabiralizumab 4 mg/kg Q2W | Phase 1a: Cabiralizumab 6 mg/kg Q2W | Phase 1a: Cabiralizumab 1mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a+1b: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W | Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W
All-Cause Mortality (participants affected / at risk) | 2/3 | 6/10 | 6/11 | 2/4 | 3/4 | 172/265 | 4/6 | 7/10
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/10 | 6/11 | 2/4 | 1/3 | 138/265 | 3/6 | 5/10
Other Adverse Events (participants affected / at risk) | 2/3 | 10/11 | 10/10 | 4/4 | 3/3 | 264/265 | 6/6 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a: Cabiralizumab 2 mg/kg Q2W (N=3) | Phase 1a: Cabiralizumab 4 mg/kg Q2W (N=10) | Phase 1a: Cabiralizumab 6 mg/kg Q2W (N=11) | Phase 1a: Cabiralizumab 1mg/kg + Nivolumab 3 mg/kg Q2W (N=4) | Phase 1a: Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W (N=3) | Phase 1a+1b: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W (N=265) | Phase 1a: Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W (N=6) | Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 40 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 11 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 9 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 8 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Necrotising granulomatous lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1a: Cabiralizumab 2 mg/kg Q2W (N=3) | Phase 1a: Cabiralizumab 4 mg/kg Q2W (N=11) | Phase 1a: Cabiralizumab 6 mg/kg Q2W (N=10) | Phase 1a: Cabiralizumab 1mg/kg + Nivolumab 3 mg/kg Q2W (N=4) | Phase 1a: Cabiralizumab 2 mg/kg + Nivolumab 3 mg/kg Q2W (N=3) | Phase 1a+1b: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q2W (N=265) | Phase 1a: Cabiralizumab 6 mg/kg + Nivolumab 3 mg/kg Q2W (N=6) | Phase 1a: Cabiralizumab 4 mg/kg + Nivolumab 3 mg/kg Q3W (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 2 | 0 | 88 | 3 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 7 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 11 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 16 | 0 | 2
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Altered visual depth perception (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 0
Episcleritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eye allergy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0
Eyelid pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Eyelid rash (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 19 | 0 | 2
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 4 | 4 | 0 | 1 | 122 | 5 | 3
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Scleritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 23 | 0 | 2
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 21 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 5 | 3 | 0 | 0 | 45 | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 13 | 0 | 0
Aphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 9 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Buccal mucosal roughening (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 69 | 4 | 2
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 1 | 69 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 19 | 2 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 14 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 25 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 6 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 8 | 1 | 0
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 0 | 0 | 87 | 1 | 4
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oesophageal irritation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 13 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 0 | 60 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 2 | 0 | 0 | 23 | 1 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 8 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 25 | 0 | 0
Decreased activity (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device malfunction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 24 | 2 | 3
Fat tissue increased (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 5 | 4 | 1 | 0 | 148 | 6 | 3
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 10 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0
Loss of control of legs (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Medical device site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 4 | 0 | 0 | 54 | 2 | 2
Pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 15 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 58 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1 | 0 | 0 | 52 | 3 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis in device (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 11 | 1 | 4
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gastrointestinal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oesophageal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 17 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scrotal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stoma site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 15 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 15 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 10 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dural tear (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye burns (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 13 | 1 | 4
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 6 | 0 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 0 | 59 | 1 | 1
Aldolase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 1 | 1 | 1 | 51 | 0 | 0
Antineutrophil cytoplasmic antibody increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 6 | 1 | 1 | 115 | 2 | 1
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Band neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 3 | 0 | 0 | 35 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 13 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 4 | 0 | 1 | 125 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 3 | 1 | 0 | 0 | 25 | 0 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 37 | 1 | 2
Blood lactic acid increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Blood urea increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Globulins increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematocrit decreased (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 0
Lipase increased (Investigations) | 0 | 3 | 1 | 1 | 1 | 49 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 3 | 0 | 1 | 0 | 20 | 0 | 0
Myoglobin blood increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thyroxine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 0
Tri-iodothyronine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 26 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1 | 0 | 68 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 27 | 5 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 14 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 29 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 20 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 39 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 13 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 44 | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 41 | 2 | 2
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 33 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 0 | 39 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Muscle oedema (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 20 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 16 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 18 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 24 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Haemorrhagic tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant lymphoid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 1 | 0 | 0 | 31 | 0 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 17 | 2 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 0 | 1 | 44 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 5 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 7 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 27 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 17 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 11 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 40 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Obsessive thoughts (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Tension (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 8 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypersthenuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urethral spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 70 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0 | 81 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 6 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 11 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 13 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 23 | 0 | 1
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 15 | 1 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0 | 26 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 14 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 6 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 15 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 10 | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 0 | 62 | 4 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0
Pseudofolliculitis barbae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1 | 68 | 2 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 37 | 1 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 1 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 12 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0
Xanthelasma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bloody discharge (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 9 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 39 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 17 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Prehypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Inclusion of multiple tumor types and several dose levels in monotherapy and combination with nivolumab limits the ability to accurately evaluate the incidence of off-target effects adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial prior to submission for publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT02526017/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT02526017/SAP_001.pdf